CLINICAL TRIAL: NCT00962572
Title: The Effects of Aggressive Patient Management on Cancer Therapy Management
Status: Withdrawn | Type: Observational
Why Stopped: Investigator decided not to pursue
Sponsor: University of Mississippi Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2008-0093
Record Dates: First submitted 2009-08-18; First posted 2009-08-20 (Estimated); Last update posted 2012-04-09 (Estimated); Status verified 2012-04

CONDITIONS: Cancer
Keywords: Outcomes; Cancer; Radiotherapy; Socio-economic
MeSH Terms: conditions — Neoplasms | interventions — Patient Care Management

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Patient management — Aggressive patient management will be implemented by a corps of "patient manager" volunteers backed by a transportation, nutrition, and social services network. The social services professionals will work with the volunteers to establish the support needed for each patient. The volunteer managers will in turn constantly monitor that such support is addressing the patient's ability to be treated. Access to sponsored housing will be coordinated. Nutritional support will be coordinated by the Dietary department and will consist of counseling, and supplements when necessary. Provision of supplemental feeding for housed patients will be arranged.

SUMMARY:
A study to see if coordinated aggressive patient management will improve patient treatment outcomes and is cost effective.

DETAILED DESCRIPTION:
This is an observational study of the effects of aggressive patient management. The records of 50 patients treated under the aggressive management plan will be matched with the records of 50 previous patients and attempts made to assess the improvement, if any, found. Statistical analysis will compare the outcomes of the study group and the matched control group for initial completion of planned therapy as per prescription, weight loss during therapy, intercurrent illness, and intercurrent hospitalizations. Long term analysis will compare the study group's outcomes (compared to expected outcomes) compared to the matched control group.

ELIGIBILITY:
Inclusion Criteria:

* live 45 minutes from treatment facility
* family income less than 200% federal poverty guideline

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: rural and minority patients who require radiation therapy
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2009-01; Primary Completion 2009-12 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
To test effects of intensive patient management on patient's compliance with referral and subsequent treatment protocol. | 1 year

SECONDARY OUTCOMES:
To test if increased compliance results in better therapy outcomes and fewer complications of the disease process as evidenced by increased survival and fewer intercurrent hospitalizations. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Michael C Baird, MD, Principal Investigator — University of Mississippi Medical Center
Locations (1):
- University of Mississippi Radiation Oncology, Jackson, Mississippi, United States